CLINICAL TRIAL: NCT01257555
Title: Evaluation of a Photopneumatic System for the Treatment of Acne
Status: Completed | Type: Observational
Sponsor: Solta Medical (Industry)
Responsible Party: Sponsor
Organization: Valeant Pharmaceuticals (Industry)
Other Study IDs: 10-116-CF-I
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Mild to Moderate Acne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Treatment Group
  Interventions: Device: Photopneumatic therapy

INTERVENTIONS:
Device: Photopneumatic therapy — Use of intense pulsed light (photo) in combination with vacuum technology (pneumatic) to treat mild to moderate acne.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of a photopneumatic therapy for the treatment of acne and concomitant symptoms associated with the disease, including erythema.

DETAILED DESCRIPTION:
The primary aims of the study will be to demonstrate the safety and efficacy of using a photopneumatic system for treatment of mild to moderate acne on the face or body - including neck, chest, and back - of up to 24 subjects. To support this clinical assessment, the affected areas to be treated will be documented at baseline, at each subsequent treatment visit (up to 6 treatments), and at one (1) month and three (3) months following final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Fitzpatrick skin type I-VI.
2. Male or female.
3. Subjects must be between 18 and 55 years of age.
4. Subjects must have mild to moderate acne (defined as 15 or more inflammatory or non-inflammatory lesions).
5. Subjects must read, understand, and sign the informed consent form.
6. Subjects must be willing and able to comply with all follow-up requirements.

Exclusion Criteria:

1. Subjects must not have active localized or systemic infections.
2. Subjects must not have a compromised ability for wound healing, such as: malnutrition, steroid use, history of collagen vascular disease (e.g. lupus, scleroderma, history of keloid scar formation), atrophic dermatitis or immunologic abnormalities such as vitiligo.
3. Subjects must not have received microdermabrasion within one (1) month prior to enrollment.
4. Subjects must not have received immunosuppressive medication(s) one (1) month prior to enrollment.
5. Subjects must not have received laser or light treatment within the last three (3) months.
6. Subjects must not have received dermabrasion, TCA peel greater than 20%, botulinum toxin type A, dermal fillers, photodynamic therapy (PDT), or cosmetic surgery within the last six (6) months .
7. Subjects must not be currently taking or have used isotretinoin (e.g. Accutane) within six (6) months prior to enrollment.
8. Subjects must agree to refrain from using cosmeceutical agents or topical agents during the course of the study, except as directed by study investigators.
9. Subjects must not have had previous ablative laser treatment.
10. Subjects must refrain from excessive sun exposure during participation in this study.
11. Subjects must not have any condition that results in photosensitivity or be taking any medication containing aminolevulinic acid (E.g. Levulan).
12. Subjects must not be a current or past smoker of cigarettes and/or cigars.
13. Subjects must not be pregnant.
14. Any condition or situation that would prevent the subject from safely completing all protocol requirements for participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All genders and ethnic backgrounds. No subjects from vulnerable categories (i.e. minors, pregnant women, etc).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Solta Medical, Hayward, California, United States